CLINICAL TRIAL: NCT03925350
Title: A Phase II Study of Niraparib in Patients With Advanced Melanoma With Genetic Homologous Recombination (HR) Mutation / Alteration
Brief Title: Efficacy and Safety Study of Niraparib in Melanoma With Genetic Homologous Recombination (HR) Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Tesaro, Inc. (Industry); Vanderbilt-Ingram Cancer Center (Other); Huntsman Cancer Institute (Other)
Responsible Party: Principal Investigator, Kevin Kim, Principal Investigator, California Pacific Medical Center Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPMC17-MEL01
Record Dates: First submitted 2019-03-15; First posted 2019-04-24 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Melanoma
Keywords: Homologous recombination (HR); Mutation; Niraparib; PARP inhibitor
MeSH Terms: conditions — Melanoma | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib (Experimental): Patients receive niraparib PO daily
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — 300 mg PO daily

SUMMARY:
This open-label phase II trial studies how well niraparib works in treating patients with advanced, metastatic melanoma with the homologous recombination (HR) pathway gene mutation / alteration. Niraparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. The trial is designed to assess the efficacy and safety of niraparib in patients with HR mutation/ alteration whose disease progressed on prior immunotherapy and/or BRAF-targeting therapy.

DETAILED DESCRIPTION:
Treatment with PARP inhibitors could represent a novel opportunity to selectively kill a subset of cancer cells with deficiencies in DNA repair pathways. For example, a tumor arising in a patient with a germline BRCA mutation (gBRCAmut) has a defective homologous recombination DNA repair pathway and would be increasingly dependent on NHEJ, alt-NHEJ, and BER for maintenance of genomic integrity. PARP inhibitors block alt-NHEJ and BER, forcing tumors with BRCA deficiencies to use the error-prone NHEJ to fix double-strand breaks. Non-BRCA deficiencies in homologous recombination DNA repair genes could also enhance tumor cell sensitivity to PARP inhibitors. The rationale for anticancer activity in a subset of non-gBRCAmut tumors is that they share distinctive DNA repair defects with gBRCAmut carriers, a phenomenon broadly described as "BRCAness." DNA repair defects can be caused by germline or somatic alterations to the homologous recombination DNA repair pathway. Homologous recombination is a complex pathway, and several genes other than BRCA1 and BRCA2 are required either to sense or repair DNA double-strand breaks via the homologous recombination pathway. Therefore, PARP inhibitors are also selectively cytotoxic for cancer cells with deficiencies in DNA repair proteins other than BRCA1 and BRCA2.

In melanoma, genetic HR mutation/ alterations are rather common. Retrospective data showed that nearly 30.5% of cutaneous melanoma harbors a mutation in at least 1 of the HR genes in their tumor. The most commonly altered gene was ARID2, followed by ARID1A, FANCA, ATM, BRCA1, ATRX and BRCA2, ATR, BRCA1 and BRIP1.

These findings provide a strong rationale to evaluate the clinical efficacy of a PARP inhibitor in patients with advanced cancers with HR mutation/alteration or HR deficiency. Therefore, the investigators propose a phase II study of niraparib in patients with advanced melanoma with genetic homologous recombination mutation/ alteration.

In this clinical study, clinical efficacy of niraparib will be evaluated by assessing an objective clinical response rate in patients with advanced, metastatic melanoma with the homologous recombination (HR) pathway gene mutation / alteration. All participating patients will receive niraparib 300 mg a day until disease progresses or they experience intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Have genetic homologous recombination (HR) mutation/ alteration including ARID1A/B, ARID2, ATM, ATR, ATRX, BARD1, BRCA1/2, BAP1, BRIP1, CHEK2, FANCD2, MRN11A, PALB2, RAD50, RAD51, RAD54B
* Disease must have progressed on the standard systemic therapies or they could not have tolerated the standard therapies.
* ECOG PS >/=1
* Have measurable metastatic disease according to RECIST 1.1
* Prior systemic cytotoxic therapy up to 1 regimens is allowed; There is no limit on the number of prior immunotherapy or targeted therapy regimens.
* All adverse events associated with prior treatment must have resolved to ≤ Grade 1 prior to day 1 of the study drug administration.

Exclusion Criteria:

* Previously treated with a PARP inhibitor
* Symptomatic brain metastasis or active brain lesions ≥6 mm size or those
* Require steroid treatment for brain lesions or leptomeningeal disease
* Systemic cancer therapy within 14 days prior to day 1 of the study drug administration
* Any major surgery ≤ 3 weeks of starting the study and patient must have recovered from any effects of any major surgery
* Investigational therapy administered ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational
* Prior radiotherapy encompassing > 20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy
* Medical history of immunocompromised condition
* Systemic treatment of another type of cancer ≤ 2 years prior to registration
* Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  ORR of niraparib in patients with advanced melanoma with genetic homologous recombination (HR) mutation/ alteration using RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS of patients with advanced melanoma with genetic HR mutation/ alteration who are treated with niraparib
overall survival (OS) | 2 years
  OS of patients with advanced melanoma with genetic HR mutation/ alteration who are treated with niraparib
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | 2 years
  Evaluation of the safety profile of niraparib treatment in patients with advanced melanoma with genetic homologous recombination (HR) mutation/ alteration

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kim, MD, Principal Investigator — California Pacific Medical Center
Locations (1):
- California Pacific Medical Center Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim KB, Desprez PY, de Semir D, Woo RWL, Sharma A, Jones R, Caressi C, Nosrati M, Janiczek E, Rivera Penafiel J, Kashani-Sabet M. Phase II Study of Niraparib in Patients With Advanced Melanoma With Homologous Recombination Pathway Gene Mutations. JCO Precis Oncol. 2025 May;9:e2400658. doi: 10.1200/PO-24-00658. Epub 2025 May 15. PMID 40373259